CLINICAL TRIAL: NCT05260879
Title: Potential Effectiveness of the Diabetes Prevention Program in the Peri-urban Area of Bamako, Mali
Acronym: PPD-Mali
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Clinical Research Center, Mali (Other)
Collaborators: Columbia University (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020/207/CE/FMOS/FAPH; 1R21TW011736-01 (NIH)
Record Dates: First submitted 2021-12-06; First posted 2022-03-02 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individuals (Experimental): This arm is composed of diabetic or hypertensive men and women who participate without joint participation of their spouse. The intervention consists of exposing participants to bi-monthly educational sessions on diet and exercise. Participants will be organized in groups of 15 led by one community health worker (CHW) assisted by a diabetes peer educator (PE). The basic format for the group sessions will follow the pattern developed with the DPP program, beginning with a discussion of "success" stories from the past weeks before proceeding to the didactic portion of the session. The sessions will mix the didactic portions facilitated by the PE with group discussions, activities and role plays, facilitated by the CHW.
  Interventions: Behavioral: Diabetes prevention program
- Couples (Experimental): Women recruited for the couples group will be asked to invite their husbands to participate, regardless of their husband's CVD status, and men whose wives do not have CVD similarly will be asked to enroll with their wife. The intervention consists in exposing them to bi-monthly educational sessions on diet and exercise. The intervention consists in exposing participants with bi-monthly educational sessions on diet and exercise. Participants will be organized in groups of 15 to 30, led by one community health worker (CHW) assisted by a diabetes peer educator (PE). The basic format for the group sessions will follow the pattern developed with the DPP program, beginning with a discussion of "success" stories from the past weeks before proceeding to the didactic portion of the session. The sessions will mix the didactic portions facilitated by the PE with group discussions, activities and role plays, facilitated by the CHW.
  Interventions: Behavioral: Diabetes prevention program
- Comparison (No Intervention): The comparison group is composed of diabetic or hypertensive individuals who agreed to participate in the study but who will not be exposed to the sessions.

INTERVENTIONS:
Behavioral: Diabetes prevention program — Adaptation of the Centers for Disease Control and Prevention (CDC) Diabetes Prevention Program Power to Prevent for use in low income neighborhoods in Bamako, Mali
  Other Names: PPD-Mali
  Arms: Couples; Individuals

SUMMARY:
The proposed research is an innovative adaptation of the Centers for Disease Control and Prevention's (CDC) Diabetes Prevention Program "Power to Prevent" program, which will be developed and piloted in the low-income peri-urban neighborhoods of Bamako, Mali. This program is well-suited to delivery by the city's community health workers already supporting families in improving maternal and child health outcomes. First, it will use participatory research methods to engage them and community residents in making adaptations to the community health worker's guidelines and tools for recommended activities so that they are linguistically and culturally appropriate, including guidelines for food consumption using locally available foods. These adaptations will use more graphics and photographs, so they are appropriate for low-literacy participants. Second, another key innovation is the explicit orientation to couples, where only one may have a diagnosed cardiovascular disease. This adaptation will provide tools the women can use in negotiating for changes to the family's meals and her daily routine. Third, investigators will conduct a comparative effectiveness study at 6 community health centers with high rates of Cardiovascular Disease (CVD), recruiting adults recently diagnosed with diabetes or hypertension. Based on the random allocation of their community health center, participants will be assigned to one of three groups of 150 each: Couples, with at least one meeting the eligibility criteria; Individuals, men and women, both eligible; Comparison, men and women with CVD. Trained community health workers and diabetic peer educators will use the adapted Diabetes Prevention Program (DPP) materials with the Couples and Individuals groups over a period of 6 months. At the conclusion of this pilot investigators will assess the levels of adoption of recommended cardiovascular risk reduction behaviors and changes in obesity, hypertension, and diabetes control, comparing differences in outcomes between the three groups. It will enable Mali to incorporate diabetes and hypertension risk reduction into their already deployed networks of community health workers. The Malian DPP adaptation will also be suitable for Francophone West Africa, where customs and lifestyles are similar among the millions of families confronting the burdens of cardiovascular disease.

DETAILED DESCRIPTION:
Specific Aims:

Aim 1 will adapt the diet and lifestyle change modalities of the Small Steps, Big Rewards (SSBR) recommendations to the cultural and economic realities affecting women's choices in Bamako. As in other cross-national adaptations of the DPP, investigators will translate the food and exercise recommendations into equivalent recommendations using locally available foods and exercise opportunities. Study partners have already estimated the caloric and glycemic indices of the most common foods prepared in Mali, and the demonstrations and recommendations will be based on these estimations. Cultural and gender-sensitive recommendations for exercise will be similarly tailored to the urban African context, with participating women from the low-income communities ensuring the cultural appropriateness of these adaptations.

Aim 2 will develop culturally and gender-specific communication strategies for empowering low- income, low-literacy women to apply the SSBR recommendations for themselves and their families. Investigators will incorporate the tools and demonstrations for SSBR developed in Aim 1 to the refinement of the Malian adaptation SSBR-Mali group sessions. An effective approach to chronic disease management in Africa has promoted sharing adherence messages among couples, so they can better support each other in staying adherent. The preliminary work also highlights the need to explore alternative methods to help women gain the approval and support of their spouses and other family members.

Aim 3 is to assess the effectiveness of the Malian adaptation of the DPP to increase adoption of diabetes prevention practices and reduce hyperglycemia and hypertension among couples enrolling in the program, compared to those participating as individuals. Using the adaptation developed in Aim 2 the investigators will compare the effectiveness of the Malian adaptation of the SSBR in selected community health centers in peripheral low-income communities with high rates of diabetes or hypertension. Trained CHWs and diabetic peer educators will implement the program for 6 months, with assessments conducted to compare changes pre-post participation in healthy behaviors and diabetes and hypertension management outcomes with 450 participants in the intervention at 4 community health centers versus 150 comparable individuals at 2 control community centers. The analysis will focus on the comparison of effectiveness for individuals enrolled as couples where at least one has CVD versus those enrolled as individuals with CVD.

Research Plan

A. Innovation

The couple-orientation to this DPP is innovative, as all previous DPP adaptations focus on individual participants. By enrolling both members of a couple where only one of them may have diabetes or hypertension, they will both participate in group sessions and learn how they can support each other to make changes. Carefully crafted role plays will provide women with the communication tools for negotiating changes to family meals or daily activities. The adaptation will be the first which recognizes the need for materials to be appropriate for low-literacy participants, with greater use of locally prepared photographic and graphic content for group sessions, the CHW flip-chart and participant food and activity tracker materials. The participatory approach to developing the pilot study will further strengthen the skills of the University of Sciences, Techniques and Technologies of Bamako (USTTB) researchers toward shifting their research out of the clinics and into the neighborhoods, enabling them to better partner with the health ministry as they move in the direction of prevention and community-based health services.

B. Approach

1. Study Site: Mali has noncommunicable diseases mortality rates among the highest in the world and higher for women than men. In 2019, the number of adults with diabetes was estimated at 157,600 adults, with only 50,000 aware of their diabetes. Bamako, the capital city with over 2 million residents, has the highest obesity and cardiovascular disease rates. Over one in ten urban adults are diabetic, and one in four hypertensive. Between 2002 and 2013 obesity among city residents aged 15-65 rose from 10% to 16%, with obesity rates five times higher for women than men. The rates of obesity and malnutrition (low diet diversity) were higher among the less educated and in low-income, peripheral neighborhoods. Therefore, this pilot study will focus on the low-income peripheral neighborhoods of Communes I and IV, where the investigators will select the six Community Health Centers (CSCOM), Mali's primary health care centers, with the highest numbers of diabetes and hypertension diagnoses in the previous two years. Four will be randomly selected to participate in the pilot, while two will serve as comparison sites.
2. Research Strategy The adaptation of the DPP SSBR program will adhere to the principles of the trans-theoretical model for facilitating behavioral change to resistant behaviors. The group lifestyle behavior approach of the DPP program is already based on the principles of the trans-theoretical change model, with the sessions helping people move quickly from pre-contemplation to contemplation (Sessions 1 and 2), preparation (Sessions 3-6), with adoption the focus of sessions 4-9, and maintenance the focus of sessions 10-12. The role plays, demonstrations, and discussions are designed to build the confidence of women to introduce healthy eating and lifestyles to their husbands and other women in their household. To ensure that the tools and activities are appropriate for the Bamako context, participatory research methods will be used, inviting 30 community residents (12 women, 12 men and 6 CHWs) from the a CSCOM to participate in the adaptation process.

To make the sessions more culturally appropriate, including the importance of involving the other women in the household in food and cooking decisions, the investigators have added sessions on how to share the responsibility for a healthy lifestyle with the other women in the household, as well as how to gain the support of the household head and other family and friends. The sessions on eating out and reading labels have been modified to be appropriate for the types of street food and market products available in Bamako. The sessions on caloric balance have been converted to the balance in the number of portions, with an emphasis on measuring portions and ingredients used in cooking. Role plays, demonstrations, and videos of exercises have been included, complementing the group discussions already included in the DPP group approach format. With these additions the number of sessions is 15, similar to that used in other group lifestyle adaptations of the DPP Power to Prevent. The training tools were pre-tested with the community health workers of a CSCOM in Bamako, and then finalized during the training of the community health workers who will deliver the program.

After the SSBR-M sessions and tools are developed, a pilot study will be conducted to assess the potential contribution that participation might make to changes in recommended behaviors of the participants and their spouses, as well as to their level of blood sugar, blood pressure, BMI and waist circumference.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25 or more
* Diagnosed with type II diabetes or hypertension or Obesity
* Willing to commit to participate at biweekly sessions for 6 months

Exclusion Criteria:

* History of stroke or cardiac arrest
* Gestational diabetes
* Type I diabetes

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Adoption of the recommended diet and exercise behavior | Month 0 to Month 6
  Number of participant who adopt the DPP recommended diet and exercise behavior

SECONDARY OUTCOMES:
Reduction in Body Mass Index (BMI) | Month 0 to Month 6
  Number of participants with reduced BMI (Weight in Kg/Height in cm) will be combined to report in kg/cm sq x10,000
Reduction in number of participants with Hypertension | Month 0 to Month 6
  Hypertension (>=140 Systole (SS) /90Diastol)
Reduction in number of participants with hyperglycemia | Month 0 to Month 6
  Hyperglycemia (>= 8.0 HbA1c)

CONTACTS AND LOCATIONS:
Overall Officials: Seydou Doumbia, MD, PhD, Principal Investigator — USTTB
Locations (6):
- Mali (6):
  - ASACOBA, Bamako
  - Asacodjeneka, Bamako
  - ASACODOU, Bamako
  - Asacola B5, Bamako
  - Asacola Ii, Bamako
  - Asacosisou, Bamako

REFERENCES:
- [Derived] Findley SE, Doumbia L, Ba HO, Maiga B, Berethe RK, Sangare HM, Besancon S, Coumare D, Coulibaly L, Cisse H, Sidibe SY, Diallo K, M'Baye R, Simaga M, Coumare M, Goita A, Diarra B, Kante M, Sanogo F, Sarro YDS, Boukenem L, Sylla SD, Nientao I, Sangho H, Kachur SP, Doumbia S. A Hybrid Effectiveness-Implementation Trial of the 'Power To Prevent Diabetes Program' in Bamako, Mali. Glob Implement Res Appl. 2026 Jan 8:10.1007/s43477-025-00199-x. doi: 10.1007/s43477-025-00199-x. Online ahead of print. PMID 41647680